CLINICAL TRIAL: NCT06692088
Title: "Longitudinal Analysis of Amylin Levels in Migraine Patients Undergoing an Anti- CGRP/CGRPr Treatment"
Status: Not yet recruiting | Type: Observational
Sponsor: Fundación Marques de Valdecilla (Other)
Collaborators: Hospital Universitario MarquÃ©s de Valdecilla (Unknown); Instituto de InvestigaciÃ³n MarquÃ©s de Valdecilla (Unknown); Clinica Universidad de Navarra, Universidad de Navarra (Other); FundaciÃ³n Marques de Valdecilla (Unknown)
Responsible Party: Principal Investigator, Gabriel Garate, Ph.D, Carlos III Health Institute
Other Study IDs: PMP22/001358; Not Yet (Other Grant/Funding Number: International Headache Society)
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: High Frequency Episodic Migraine and Chronic Migraine
Keywords: Migraine; Amylin; Anti-CGRP/CGRPr monoclonal antibodies
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples will be obtained from blood extractions of peripheral circulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Migraine: Patients diagnosed with either high frecuancy episodic or chronic migraine and prescribed with anti-CGRP/CGRPr monoclonal antibodies without having started their treatment.
- Healthy controls: Subjects without history of migraine or any other primary headache.

SUMMARY:
Migraine, a complex and multifaceted disorder, remains only partially understood, with therapeutic strategies often limited by individual variability in response. While targeting calcitonin gene-related peptide (CGRP) has transformed migraine management, approximately half of patients with therapies targeting the CGRP pathway experience insufficient relief, suggesting other molecular players in migraine pathophysiology may be overlooked. Emerging evidence highlights amylin, a peptide of the calcitonin family, as a promising candidate with potential mechanistic overlap with CGRP. Canonical receptor of amylin is known to interact with CGRP, and both peptides are expressed in structures relevant to migraine. Preliminary clinical findings suggest that amylin might be involved in migraine pathophysiology by developing attacks and contributing to chronification of the condition; however, its exact impact and clinical relevance remain unverified.

This prospective, monocentric, cross-sectional pilot study aims to deepen our understanding of the role of amylin in chronic migraine and anti-CGRP treatment outcomes. Specifically, we will (1) measure baseline interictal serum amylin levels in chronic migraine patients receiving anti-CGRP or CGRP receptor monoclonal antibody (mAb) therapy and a group of controls matched by sex and age, (2) monitor changes in amylin levels after six months of treatment, and (3) assess the correlation between amylin levels and clinical outcomes.

We hypothesize that baseline amylin levels will be elevated in migraine patients and will normalize following effective treatment, aligning with improved clinical outcomes. Conversely, persistently elevated amylin levels may correlate with poorer response rates, potentially explaining the variability of treatment outcome found in the migraine population.

DETAILED DESCRIPTION:
While the discovery of calcitonin gene-related peptide (CGRP) and its role in migraine has offered important insights into the condition and currently offers an effective pharmacological target for many patients, it fails to explain the variability of this complex disorder (Ashina et al. 2021). Unsurprisingly, some patients do not benefit from the use of anti-CGRP therapies (Caronna et al. 2024), gepants and/or monoclonal antibodies (mAb), raising the question of what else we are missing in the migraine pathophysiology, and whether other targets could complement the current treatment options (Rees et al. 2022).

In this context, different research studies have pointed to a wide range of candidates, though results remain inconclusive (Silvestro et al. 2023). One of the most promising candidates is amylin, a 37-amino acid peptide (Hay 2017), which is a member of the calcitonin family, where CGRP is also found. In fact, the existence of a relationship between CGRP and amylin is well documented, as these two molecules show some promiscuity with each other's receptors. Specifically, the receptor for amylin shares the same affinity for its canonical ligand (CGRPr) as it has for CGRP (Hay et al. 2018). Besides the signalling overlap found between CGRP and amylin there are some other features that indicate a possible implication of this endocrine peptide in migraine. The expression of both ligand and receptor, although it is primarily found in the pancreas, where amylin develops its main function as glucose-lowering hormone (Lutz 2005), is not limited to it. Amylin and its receptor are also expressed in migraine relevant sites, including sensory neurons (Mulder et al. 1995) and the trigeminovascular system (Hendrikse et al. 2019). Moreover, amylin is also implicated in pain processing, a key feature of migraine pathophysiology, despite its precise role within pain mechanisms is poorly understood (Hay et al. 2017). Overall, the knowledge we currently got about amylin, its overlapping signalling, locations, and functions, clearly points to a degree of implication for the molecule or its receptor in the pathophysiology of the migraine attack, although its precise involvement remains undescribed and still has a lot of questions remaining to be answered.

Over the last few years, efforts have been made to advance our knowledge about the relevance of amylin receptor-dependent pathways in migraine (Russo & Hay 2023). Provocation studies in mice support a role of the peptide in inducing cutaneous sensitivity and photophobia (De Logu et al. 2019; Ghanizada et al. 2021), providing proof of principle that amylin and CGRP might have overlapping functional roles. When we focus on humans, a Danish clinical trial study found that the infusion of pramlintide, an amylin receptor agonist used in clinical practise for the treatment of diabetes, in a group of patients diagnosed with migraine without aura provoked immediate headache and migraine-like headache in a very similar proportion and characteristics to the ones produced by the infusion of CGRP in the same subjects (Ghanizada et al. 2021). It also showed that despite a third of patients who developed migraine-like attacks did so with both molecules there was an important proportion who were only sensitive to either amylin or CGRP, but this observation requires further investigation.

Complementary to these data, there is a case-control study which investigated the interictal levels of amylin and CGRP in a group of patients with episodic or chronic migraine (Irimia et al. 2021). The research found both peptide concentrations were increased only in the chronic migraine group when compared to controls and patients with episodic migraine. Although the main aim of this research was to evaluate the usefulness of amylin as a biomarker for chronic migraine it raised the question of whether amylin could be playing a role in migraine chronification, similarly to what has been hypothesized with CGRP (Torres-Ferrús et al. 2023). To this date, there is not any additional study which has confirmed/refuted these findings, so their conclusions should be taken carefully.

Lastly, we have the evidence coming from studies evaluating the impact of mAbs targeting the free ligand or the CGRP. Real word data reveal that these two different approaches have almost identical rates of efficacy (Haghdoost et al. 2023). This initially came as a surprise as the different targeting of these therapeutic agents could provide different outcome rates. Blocking CGRP itself acts on both the canonical receptor but also on the amylin receptor, whose signalling would now solely depend on the amylin itself. On the other side, targeting the classical receptor of CGRP theoretically would still allow the interaction of the ligand with the amylin receptor, although recent studies have found that erenumab also interacts with this receptor, but with a lesser selectivity than it has with CGRPr (Garelja et al. 2024). The question of whether this newly described interaction has a meaningful effect on amylin receptor signalling is still a mystery. Moreover, several studies have evaluated the concentrations of CGRP in chronic migraine during the course of mAb therapies (Alpuente et al. 2022; Raffaelli et al. 2023), and it has been showed a link between higher basal interictal concentrations of alpha-CGRP and a tendency to have a better response to the therapies independently of their mechanism of action (Alpuente et al. 2022; Gárate et al. 2023), but there is a lack of explanation specifically linked to the CGRP-levels to why almost half of the patients do not benefit from the medication. Finally, not all patients have elevated levels of CGRP (Gárate et al. 2024), as the large dispersion of data found across studies found proves, and taking all the data together, a plausible explanation would be that some of the migraine attacks, if not the migraine condition itself, could be CGRP-independent in some of the patients, and consequently depend on other molecules.

To conclude, amylin is, due to its overlapping properties with CGRP and the recently published data, one of the most promising candidates to become the second molecule able to explain the heterogeneity found in migraine. However, a lot of information remain to be understood before potentially offer a new therapeutic target option or act as biomarker for this condition. This process will undoubtedly require research, as it is the only way to expand our knowledge and achieve a successful translation for the amylin from the bench to the clinic.

SPECIFIC AIMS AND HYPOTHESIS

Our specific aims are the following:

Evaluate the interictal circulating levels of amylin in serum within the context of an anti-CGRP/CGRPr mAb treatment.

Analyse the evolution of these concentrations after the first 6 months of treatment.

Assess the possible correlation of the concentrations with clinical parameters of our patients.

Compare the results at basal and at 6 months after initiation of treatment with a group of controls.

We hypothesized that basal levels of amylin will be elevated compared to control group, as described previously, that these concentrations will vary after 6 months of treatment these concentrations will vary, and their evolution will correlate with clinical and/or response variables.

METHODS

This is a prospective, monocentric, cross sectional, pilot study.

Adequacy of the group

The Headache Unit of the University Hospital Marqués de Valdecilla has a proven record of migraine management and currently has more than 400 patients with an active anti-CGRP/r mAb treatment. Furthermore, our group is pioneer in the measurement of neuropeptides, such as CGRP, VIP or PACAP, with a proven track of multiple publications on this topic among top tier journals (Cernuda-Morollón et al. 2014; Riesco et al. 2017; Pérez-Pereda et al. 2020; Irimia et al. 2021; Gárate et al. 2023; Gárate et al. 2024). Altogether, we believe we have the human resources and know-how and experience to carry out a project of the defined characteristics.

Patients and controls

Patients fulfilling chronic migraine criteria and prescribed with these therapeutic agents will be asked to enrol in this study. Clinical data will be prospectively recorded from the moment of joining the study as well as previous relevant clinical data, which will be collected by interviewing the patient and by reviewing their clinical history. The control group will consist in subjects with absence of migraine history or any other kind of primary headache that will be paired to the migraine group by sex and age. These will be recruited from workers from the hospital and their families who altruistically volunteer to participate.

Sample size

Based on the results from Irimia et al 2021 we calculated that with an expected difference means of 35%, an alpha equal to 0.01 and a power of 80% we had to include a minimum of 61 participants per group.

Sample collection, processing and storage

All blood samples will be extracted by nurses from the Headache Unit in our hospital facilities. Following the guidelines for analysing CGRP in serum set by a recent article (Gárate et al. 2024), the standard conditions to perform the sampling are: (1) at least 12 hours fasting; (2) blood from cubital vein extracted between 9-12 am; (3) at least 24 hours of free headache period; (4) no use of any kind of analgesic medication in the previous 24 hours. Additionally, the patients with migraine cannot have taken any symptomatic treatment to abort their migraine attack in the previous 24 hours. The concomitant use of preventives apart from the recently prescribed anti-CGRP/r mAb is allowed.

All samples will be allowed to clot, immediately centrifuged, aliquoted and stored at 4oC up to 6 hours, until serum is finally transferred into a freezer at -80oC. No sample will be stored more than 4 months before being analysed.

Molecular determinations

Serum amylin concentrations will be determined by a validated fluorescent sandwich ELISA specifically designed for the detection of the active form of the peptide and without any remarkable cross reactivity for analogues (<1%) which has already been employed in previous works (Irimia et al. 2021).

Data analysis

The statistical analysis will be performed with specific software, GraphPad Prism and SPSS. Serum amylin concentrations will be compared between controls and the migraine group as well as within the migraine group throughout the treatment. Analysis will also include the evaluation of possible correlations between clinical/treatment variables and the levels of the neuropeptide and the comparison among subgroups of patients with migraine based on post-hoc classifications.

REFERENCES

Alpuente, A., Gallardo, V. J., Asskour, L., Caronna, E., Torres-Ferrus, M., & Pozo-Rosich, P. (2022). Salivary CGRP and Erenumab Treatment Response: Towards Precision Medicine in Migraine. Annals of Neurology, 92(5), 846-859. https://doi.org/10.1002/ana.26472

Ashina, M., Terwindt, G. M., Al-Karagholi, M. A. M., de Boer, I., Lee, M. J., Hay, D. L., Schulte, L. H., Hadjikhani, N., Sinclair, A. J., Ashina, H., Schwedt, T. J., & Goadsby, P. J. (2021). Migraine: disease characterisation, biomarkers, and precision medicine. In The Lancet (Vol. 397, Issue 10283, pp. 1496-1504). Elsevier B.V. https://doi.org/10.1016/S0140-6736(20)32162-0

Caronna, E., Gallardo, V. J., Egeo, G., Vázquez, M. M., Castellanos, C. N., Membrilla, J. A., Vaghi, G., Rodríguez-Montolio, J., Fabregat Fabra, N., Sánchez-Caballero, F., Jaimes Sánchez, A., Muñoz-Vendrell, A., Oliveira, R., Gárate, G., González-Osorio, Y., Guisado-Alonso, D., Ornello, R., Thunstedt, C., Fernández-Lázaro, I., … EUREkA study group. (2024). Redefining migraine prevention: early treatment with anti-CGRP monoclonal antibodies enhances response in the real world. Journal of Neurology, Neurosurgery, and Psychiatry. https://doi.org/10.1136/jnnp-2023-333295

Cernuda-Morollón, E., Mart\'\inez-Camblor, P., Ramón, C., Larrosa, D., Serrano-Pertierra, E., & Pascual, J. (2014). CGRP and VIP levels as predictors of efficacy of Onabotulinumtoxin type A in chronic migraine. Headache, 54(6), 987-995.

de Logu, F., Landini, L., Janal, M. N., Li Puma, S., de Cesaris, F., Geppetti, P., & Nassini, R. (2019). Migraine-provoking substances evoke periorbital allodynia in mice. Journal of Headache and Pain, 20(1). https://doi.org/10.1186/s10194-019-0968-1

Debbie Hay, C. L., Hay, D. L., Garelja, M. L., Poyner, D. R., & Walker, C. S. (2018). Update on the pharmacology of calcitonin/CGRP family of peptides: IUPHAR Review 25. British Journal of Pharmacology, 175(3), 3-17. https://doi.org/10.1111/bph.13878/full

Gárate, G., González-Quintanilla, V., González, A., Pascual, M., Pérez-Pereda, S., Madera, J., & Pascual, J. (2023). Serum Alpha and Beta-CGRP Levels in Chronic Migraine Patients Before and After Monoclonal Antibodies Against CGRP or its Receptor. Annals of Neurology, 94(2). https://doi.org/10.1002/ana.26658

Gárate, G., Pascual, J., Pascual-Mato, M., Madera, J., Martín, M. M. S., & González-Quintanilla, V. (2024). Untangling the mess of CGRP levels as a migraine biomarker: an in-depth literature review and analysis of our experimental experience. Journal of Headache and Pain, 25(1). https://doi.org/10.1186/s10194-024-01769-4

Garelja, M. L., Alexander, T. I., Bennie, A., Nimick, M., Petersen, J., Walker, C. S., & Hay, D. L. (2024). Pharmacological characterisation of erenumab, Aimovig, at two calcitonin gene-related peptide responsive receptors. British Journal of Pharmacology, 181(1), 142-161. https://doi.org/10.1111/bph.16218

Ghanizada, H., Al-Karagholi, M. A. M., Walker, C. S., Arngrim, N., Rees, T., Petersen, J., Siow, A., Mørch-Rasmussen, M., Tan, S., O'Carroll, S. J., Harris, P., Skovgaard, L. T., Jørgensen, N. R., Brimble, M., Waite, J. S., Rea, B. J., Sowers, L. P., Russo, A. F., Hay, D. L., & Ashina, M. (2021). Amylin Analog Pramlintide Induces Migraine-like Attacks in Patients. Annals of Neurology, 89(6), 1157-1171. https://doi.org/10.1002/ana.26072

Haghdoost, F., Puledda, F., Garcia-Azorin, D., Huessler, E. M., Messina, R., & Pozo-Rosich, P. (2023). Evaluating the efficacy of CGRP mAbs and gepants for the preventive treatment of migraine: A systematic review and network meta-analysis of phase 3 randomised controlled trials. In Cephalalgia (Vol. 43, Issue 4). SAGE Publications Ltd. https://doi.org/10.1177/03331024231159366

Hay, D. L. (2017). Amylin. Headache, 57, 89-96. https://doi.org/10.1111/head.13077

Hendrikse, E. R., Bower, R. L., Hay, D. L., & Walker, C. S. (2019). Molecular studies of CGRP and the CGRP family of peptides in the central nervous system. In Cephalalgia (Vol. 39, Issue 3, pp. 403-419). SAGE Publications Ltd. https://doi.org/10.1177/0333102418765787

Irimia, P., Martínez-Valbuena, I., Mínguez-Olaondo, A., Domínguez-Vivero, C., Sánchez-Arias, J. A., Martínez-Vila, E., Luquin, M. R., & Leira, R. (2021). Interictal amylin levels in chronic migraine patients: A case-control study. Cephalalgia, 41(5), 604-612. https://doi.org/10.1177/0333102420977106

Lutz, T. A. (2005). Pancreatic Amylin as a Centrally Acting Satiating Hormone. In Current Drug Targets (Vol. 6).

Mulder, H., Leckstriim, A., Uddman, R., Ekblad, E., ' Per, W. :, & Sundiet-', F. (1995). Islet Amyloid Polypeptide (Amylin) Is Expressed in Sensory Neurons. In The Journal of Neuroscience (Vol. 75, Issue 11).

Pérez-Pereda, S., Toriello-Suárez, M., Ocejo-Vinyals, G., Guiral-Foz, S., Castillo-Obeso, J., Montes-Gómez, S., Martínez-Nieto, R. M., Iglesias, F., González-Quintanilla, V., & Oterino, A. (2020). Serum CGRP, VIP, and PACAP usefulness in migraine: a case-control study in chronic migraine patients in real clinical practice. Molecular Biology Reports, 47(9), 7125-7138. https://doi.org/10.1007/s11033-020-05781-0

Raffaelli, B., Terhart, M., Fitzek, M. P., Lange, K. S., Mecklenburg, J., Overeem, L. H., Siebert, A., Storch, E., & Reuter, U. (2023). Change of CGRP Plasma Concentrations in Migraine after Discontinuation of CGRP-(Receptor) Monoclonal Antibodies. Pharmaceutics, 15(1), 1-9. https://doi.org/10.3390/pharmaceutics15010293

Rees, T. A., Hendrikse, E. R., & Walker, C. S. (2022). Beyond CGRP : The calcitonin peptide family as targets for migraine and pain. British Journal of Pharmacology, 179, 381-398. https://doi.org/10.1111/bph.15605

Riesco, N., Cernuda-Morollón, E., Martínez-Camblor, P., Pérez-Alvarez, A. I., Verano, L., García-Cabo, C., Serrano-Pertierra, E., & Pascual, J. (2017). Relationship between serum levels of VIP, but not of CGRP, and cranial autonomic parasympathetic symptoms: A study in chronic migraine patients. Cephalalgia, 37(9), 823-827. https://doi.org/10.1177/0333102416653232

Russo, A. F., & Hay, D. L. (2023). CGRP physiology, pharmacology, and therapeutic targets: migraine and beyond. In Physiological reviews (Vol. 103, Issue 2, pp. 1565-1644). NLM (Medline). https://doi.org/10.1152/physrev.00059.2021

Silvestro, M., Iannone, L. F., Orologio, I., Tessitore, A., Tedeschi, G., Geppetti, P., & Russo, A. (2023). Migraine Treatment: Towards New Pharmacological Targets. In International Journal of Molecular Sciences (Vol. 24, Issue 15). Multidisciplinary Digital Publishing Institute (MDPI). https://doi.org/10.3390/ijms241512268

Torres-Ferrús, M., Ursitti, F., Alpuente-Ruiz, A., Brunello, F., Chiappino, D., de Vries, T., di Marco, S., Ferlisi, S., Guerritore, L., Gonzalez-Garcia, N., Gonzalez-Martinez, A., Khutorov, D., Kritsilis, M., Kyrou, A., Makeeva, T., Minguez-Olaondo, A., Pilati, L., Serrien, A., Tsurkalenko, O., … Lampl, C. (2020). From transformation to chronification of migraine: Pathophysiological and clinical aspects. In Journal of Headache and Pain (Vol. 21, Issue 1). BioMed Central Ltd. https://doi.org/10.1186/s10194-020-01111-8

ELIGIBILITY:
Inclusion Criteria for patients:

* Diagnosed with either: a) High Frequency Episodic Migraine or b) Chronic Migraine
* Prescribed with anti-CGRP/CGRPr monoclonal antibodies whi have not yet started his/her treatment.

Inclusion Criteria for healthy volunteers:

* No history or migraine or any other kind of headache.
* Daily consumption of any kind of analgesic treatment.

Exclusion Criteria:

* Younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Our study population are patients diagnosed with either High High Frequency Episodic Migraine or Chronic Migraine who fulfil the criteria set by our institution to be prescribed an anti-CGRP/CGRPr monoclonal antibody by our body of neurology specialist.
Sampling Method: Non-Probability Sample
Enrollment: 216 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Circulating concentrations of Amylyn | Up to 6 months
  Levels of amylin across the different time points.

OTHER OUTCOMES:
Evolution of Monthly Migraine Days (MMDs) | 6 months
  Evolution of MMDs from basal to the 6th month of treatment
Evolution of Monthly Headache Days (MHDs) | 6 months
  Evolution of MHDs from basal to the 6th month of treatment
Evolution of medication intake | 6 months
  Evolution of mediation intake from basal to the 6th month of treatment

IPD SHARING:
Plan to Share IPD: Undecided